CLINICAL TRIAL: NCT03240861
Title: Adoptive Transfer of NY-ESO-1 TCR Engineered Peripheral Blood Mononuclear Cells (PBMC) and Peripheral Blood Stem Cells (PBSC) After a Myeloablative Conditioning Regimen, With Administration of Interleukin-2, in Patients With Advanced Malignancies
Brief Title: Genetically Engineered PBMC and PBSC Expressing NY-ESO-1 TCR After a Myeloablative Conditioning Regimen to Treat Patients With Advanced Cancer
Acronym: NYESO SCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-000511; NCI-2017-00896 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Ribas NYESO SCT Cancer
Record Dates: First submitted 2017-06-22; First posted 2017-08-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: HLA-A*0201 Positive Cells Present; Locally Advanced Malignant Neoplasm; NY-ESO-1 Positive; Unresectable Malignant Neoplasm; Sarcoma
Keywords: T cells; stem cells; gene therapy; NYESO; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — 9-(4-fluoro-3-hydroxymethylbutyl)guanine; aldesleukin; Busulfan; Cell- and Tissue-Based Therapy; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Leukapheresis; plerixafor; ferric pyrophosphate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Genetically engineered PBMC and PBSC) (Experimental): G-CSF AND PLERIXAFOR MOBILIZED LEUKAPHERESIS: Between 6 months and 3 weeks before infusion of cells, patients undergo G-CSF and plerixafor mobilization of CD34+ peripheral blood stem cells. Patients receive G-CSF SC on mobilization days 1-8 and plerixafor SC on mobilization days 4-7. Patients also undergo an unmobilized leukapheresis on day -5 before infusion of cells.
  CHEMOTHERAPY CONDITIONING REGIMEN: Patients receive busulfan IV on days -4 to -2 and fludarabine IV over 30 minutes on days -3 to -2.
  Patients receive LV-NYESO TCR/sr39TK PBSC IV on day 0, and after approximately 24 hours, patients receive RV-NYESO TCR PBMC IV on day 1. Beginning on day 2, patients receive aldesleukin SC BID for up to 7 days. Patients undergo blood collection for safety and immune monitoring on days 0, 1, 3, 5, 7, 14, 30, 60, 90, and 120. Patients receive 18F-FHBG IV, and after 1 hour, undergo PET/CT on days 25 and 120.
  Interventions: Other: 18F-FHBG; Biological: Aldesleukin; Drug: Busulfan; Biological: Cellular Therapy; Procedure: Computed Tomography; Biological: Filgrastim; Drug: Fludarabine; Procedure: Leukapheresis; Drug: Plerixafor; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: 18F-FHBG — Given IV
  Other Names: Reporter Probe 18F-FHBG
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Biological: Cellular Therapy — Given LV-NYESO TCR/sr39TK PBSC IV and RV-NYESO TCR PBMC IV
  Other Names: Cell Therapy
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; Filgrastim-sndz; G-CSF; Granix; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim; Zarxio
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I clinical trial evaluates the safety and feasibility of administering NY-ESO-1 TCR (T cell receptor)engineered peripheral blood mononuclear cells (PBMC) and peripheral blood stem cells (PBSC) after a myeloablative conditioning regimen to treat patients with cancer that has spread to other parts of the body. The conditioning chemotherapy makes room in the patient?s bone marrow for new blood cells (PBMC) and blood-forming cells (stem cells) to grow. Giving NY-ESO-1 TCR PBMC and stem cells after the conditioning chemotherapy is intended to replace the immune system with new immune cells that have been redirected to attack and kill the cancer cells and thereby improve immune system function against cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of administering the combination of autologous peripheral blood mononuclear cells (PBMC) and CD34+ peripheral blood stem cells (PBSC) following a reduced intensity conditioning regimen, both of which have been genetically modified to express NY-ESO-1 TCR.

SECONDARY OBJECTIVES:

I. To determine the feasibility of delivering the combination of TCR transduced autologous PBMC and CD34+ PBSC to patients.

II. To determine the persistence of NY-ESO-1 TCR transduced PBMC and the progeny of TCR transduced PBSC in serial peripheral blood samples.

III. Objective response rate (ORR).

EXPLORATORY OBJECTIVE:

I. To explore the use of positron emission tomography (PET)-based imaging using the PET tracer 9-4-[18F]fluoro-3-(hydroxymethyl)butylguanine ([18F]FHBG) with the goal of determining whether the adoptively transferred NY-ESO-1 TCR transduced PBSC home to bone marrow, differentiate into T cells and expand in secondary lymphoid organs and tumor deposits.

OUTLINE:

G-CSF AND PLERIXAFOR MOBILIZED LEUKAPHERESIS: Between 6 months and 3 weeks before infusion of cells, patients undergo G-CSF and plerixafor mobilization of CD34+ peripheral blood stem cells. Patients receive G-CSF subcutaneously (SC) on mobilization days 1-8 and plerixafor SC on mobilization days 4-7, during mobilization, patients will undergo mobilized leukapheresis to obtain PBSC. Patients also undergo an unmobilized leukapheresis on day -5 before infusion of cells in order to obtain PBMC.

CHEMOTHERAPY CONDITIONING REGIMEN: Patients receive busulfan intravenously (IV) on days -4 to -2 and fludarabine IV over 30 minutes on days -3 to -2.

Patients receive LV-NYESO TCR/sr39TK PBSC IV on day 0, and after approximately 24 hours, patients receive RV-NYESO TCR PBMC IV on day 1. Beginning on day 2, patients receive aldesleukin (interleukin-2 (IL) or IL-2) SC twice daily (BID) for up to 7 days. Patients undergo blood collection for safety and immune monitoring on days 0, 1, 3, 5, 7, 14, 30, 60, 90, and 120. Patients receive the PET tracer 18F-FHBG IV, and after 1 hour, undergo PET/computed tomography (CT) on days 25 and 120.

After completion of study treatment, patients are followed up every 2-3 months for 2 years, every 6 months for 5 years, and annually for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or locally advanced unresectable cancers for which no alternative therapies with proven survival advantage are available
* NY-ESO-1 positive malignancy by immunohistochemistry (IHC) utilizing commercially available NY-ESO-1 antibodies
* HLA-A*0201 (HLA-A2.1) positivity by molecular subtyping
* Age greater than or equal to 16 years old; if patients 16-17 years old are enrolled in the trial, they will only be enrolled after 3 patients >= 18 years old have been treated, and the treatment has been shown to be safe
* A minimum of one measurable lesion defined as:

  * Meeting the criteria for measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)
  * Skin lesion(s) selected as non-completely biopsied target lesion(s) that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Adequate bone marrow and major organ function to undergo a PBSC transplant determined within 30-60 days prior to enrollment using standard phase 1 criteria for organ function defined as:

  * Absolute neutrophil count (ANC) >= 1.5 x 10^9 cells/L
  * Platelets >= 100 x 10^9/L
  * Hemoglobin >= 9 g/dL
  * Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x ULN (upper limit of normal) (=< 5 x ULN, if documented liver metastases are present)
  * Total bilirubin =< 2 x ULN (except patients with documented Gilbert?s syndrome)
  * Creatinine < 2 mg/dl (or a glomerular filtration rate > 60)
* Must be willing and able to accept at least three leukapheresis procedures
* Must be willing and able to undergo three research PET scans
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Inability to purify >= 2.5 x 10^6 CD34-enriched cells/kg of patient weight from the pooled G-CSF mobilized leukapheresis products
* Previously known hypersensitivity to any of the agents used in this study; known sensitivity to busulfan or fludarabine
* Received systemic treatment for cancer, including immunotherapy, within 28 days prior to initiation of conditioning chemotherapy administration within this protocol
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed)
* Human immunodeficiency virus (HIV) seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lymphodepletion; if there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the chemotherapy conditioning regimen and supportive treatments; if there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Known clinically active brain metastases; prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment and there are no neurological signs of potential brain metastases
* Pregnancy or breast-feeding; female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and for 6 months afterwards; all female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 14 days from starting the conditioning chemotherapy; the definition of effective contraception will be based on the judgment of the study investigators
* Since IL-2 is administered following cell infusion:

  * Patients will be excluded if they have a history of clinically significant electrocardiogram (ECG) abnormalities, symptoms of cardiac ischemia with evidence of ischemia on a cardiac stress test (stress thallium, stress multigated acquisition [MUGA], dobutamine echocardiogram or other stress test)
  * Similarly, patients with a baseline left ventricular ejection fraction (LVEF) < 45% will be excluded.
  * Patients with ECG results of any conduction delays (PR interval > 200 ms, corrected QT [QTC] > 480 ms), sinus bradycardia (resting heart rate < 50 beats per minute), sinus tachycardia (heart rate >120 beats per minute) will be evaluated by a cardiologist prior to starting the trial; patients with any arrhythmias, including atrial fibrillation/atrial flutter, excessive ectopy (defined as > 20 premature ventricular contractions [PVCs] per minute), ventricular tachycardia or 3rd degree heart block will be excluded from the study unless cleared by a cardiologist
  * Patients with pulmonary function test abnormalities as evidenced by a (forced expiratory volume 1 [FEV1]/forced vital capacity [FVC ] < 70% of predicted for normality will be excluded
* Bone marrow involvement based on PET/CT scan at screening
* Active or recent herpes simplex virus (HSV) infection or cytomegalovirus (CMV) based on symptoms with positive swab culture and/or positive IgM (immunoglobulin M) screening
* Liver metastases with no other metastatic sites

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | Up to 90 days
  Safety will be assessed by monitoring and recording potential adverse effects of the treatment using the Common Toxicity Criteria at each study visit. Subjects will be monitored by medical histories, physical examinations and blood studies to detect potential toxicities from the treatment. If there are no dose limiting toxicities observed, the cohort will be expanded to 12 subjects. If 1/3 are observed, up to 6 subjects will be recruited. If less than 2/6 are observed, the cohort will be expanded to a total of 12 subjects. If a dose limiting toxicity is observed in 2 or more of 6 subjects, the

SECONDARY OUTCOMES:
Detection of replication competent retrovirus and replication competent lentivirus | Up to 12 months post cell administration
  Will be assessed by polymerase chain reaction.
Duration of overall complete response | From the time measurement criteria has been first met for complete response until the first date that recurrent or progressive disease is objectively documented, assessed up to 15 years
  Will evaluate duration of overall complete response.
Duration of overall response | From the time measurement criteria is met for complete response/partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 15 years
  Will evaluate duration of overall response.
Persistence of transduced T cells | Time Frame: Up to 2 years after transgenic cell adoptive transfer
  Analysis will be performed using immune monitoring techniques. The number of days until the percentage of cells expressing both NYESO-
  1 TCR and CD3 drops below the baseline percentage.
Engraftment and persistence of transduced progeny T cells | Time Frame: Up to 2 years after transgenic cell adoptive transfer
  Analysis will be performed using immune monitoring techniques. The number of days until the vector copy number in the progeny T cells is undetectable.
Engraftment and persistence of transduced T cells and progeny T cells | Time Frame: Up to 2 years after transgenic cell adoptive transfer
  Analysis will be performed both using immune monitoring and molecular techniques.
  The number of days until the vector copy number in the T cells is undetectable.
Feasibility of generation NY-ESO-1 TCR transgenic T cells and NY-ESO-1 TCR/sr39TK transgenic stem cells that meet the lot release criteria | Time Frame: Up to 1 month after transgenic cell adoptive transfer
  Feasibility of manufacturing will be assessed as:
  The number of manufacturing products meeting the lot release criteria after an acceptable number of CD34+ cells have been obtained.
Immunological monitoring will consist primarily of quantifying T cells bearing surface NY-ESO-1 TCR | Up to 15 years
  Will be assessed by NY-ESO-1126-157/MHC (major histocompatibility complex) dextramer analysis. Functional assays like enzyme-linked immunosorbent assay, intracellular cytokine staining, and/or multicytokine array assays will complement the results. Immunological assays will be compared between 1) pre-infusion peripheral blood mononuclear cells and peripheral blood stem cells, 2) an aliquot of the engineered peripheral blood lymphocytes and stem cells at the time of infusion and 3) cells recovered from patients? peripheral blood after adoptive transfer.
Objective response | Up to 15 years
  Potential objective responses to this combinatorial immunotherapy will be recorded following Response Evaluation Criteria in Solid Tumors version 1.1 criteria.
Persistence of TCR gene transduced cells | Up to 15 years
  Will be assessed by semi quantitative deoxyribonucleic acid-polymerase chain reaction using primers specific for vector sequence.
Time to disease progression | Time from the date of cell infusion (day 0) to the date of progressive disease first documented, or death whichever occurs first, assessed up to 15 years
  Will evaluate length of time until disease progression.

OTHER OUTCOMES:
Regional uptake of 18F-FHBG within metastatic tumor sites and secondary lymphoid organs | Up to 15 years
  Will be quantified by standardized uptake values normalized to the body weight of the patient. As an internal quality control, standardized uptake values will also be determined for several normal organs, such as muscle, liver and lungs. These measurements will allow us to identify technical problems in the standardized uptake value calculations, such as partially paravenous tracer administration. Findings from non-invasive positron emission tomography imaging will be compared with results from immune monitoring assays in blood samples at different intervals after NY-ESO-1 TCR cell transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Scott Nowicki, M.D., Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Nowicki TS, Deen NNA, Peters CW, Comin-Anduix B, Medina E, Puig-Saus C, Carretero IB, Kaplan-Lefko P, Macabali MH, Garcilazo IP, Chen D, Pang J, Berent-Maoz B, Haile S, Rodriguez J, Kawakami M, Kidd CK, Champhekar A, Carlucci G, Vega-Crespo A, Chmielowski B, Singh A, Federman N, Schiller GM, Larson SJ, Allen-Auerbach M, Klomhaus AM, Zack J, Baltimore D, Yang L, Kohn DB, Witte ON, Ribas A. Human cancer-targeted immunity via transgenic hematopoietic stem cell progeny. Nat Commun. 2025 Jul 1;16(1):5599. doi: 10.1038/s41467-025-60816-z. PMID 40593578